CLINICAL TRIAL: NCT07089888
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Dotinurad Compared With Allopurinol in Adult Participants With Tophaceous Gout
Brief Title: A Study of Dotinurad Versus Allopurinol in Tophaceous Gout
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crystalys Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FYU-981-CRYS-302; 2024-520207-84-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tophaceous Gout
Keywords: Tophaceous Gout; Dotinurad; Allopurinol; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Allopurinol; dotinurad

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allopurinol (Active Comparator): Participants will discontinue their allopurinol and start on study-supplied allopurinol at the same dose once a day (QD) through Week 76.
  Interventions: Drug: Allopurinol
- Dotinurad (Experimental): Participants will discontinue their allopurinol and start dotinurad 1 mg QD for first 4 weeks (Weeks 1-4), dotinurad 2 mg QD for the next 8 weeks (Weeks 5-12), and dotinurad 4 mg QD thereafter up through Week 76.
  Interventions: Drug: Dotinurad

INTERVENTIONS:
Drug: Allopurinol — Over-encapsulated tablets containing active drug substance administered orally (PO).
  Arms: Allopurinol
Drug: Dotinurad — Over-encapsulated tablets containing active drug substance administered PO.
  Arms: Dotinurad

SUMMARY:
The primary objective of this study is to evaluate the efficacy of dotinurad in lowering serum uric acid (sUA) at Week 24 compared with allopurinol in adult participants with tophaceous gout.

ELIGIBILITY:
Inclusion Criteria

1. Between 18 and 75 years of age (inclusive) at the time of signing informed consent.
2. Diagnosis of gout based on 2015 American College of Rheumatology-European Union League Against Rheumatism (ACR-EULAR) criteria for at least 1 year.
3. Has ≥1 measurable tophus on the hands/wrists and/or feet/ankles between Screening and Day 1. A measurable tophus is defined as ≥5 mm and ≤30 mm in the longest diameter.
4. sUA level ≥5.0 mg/dL at Screening Visit 1 (Day -35 Visit) and Screening Visit 2 (Day -7 Visit).
5. Female participants of childbearing potential must have a negative serum pregnancy test at Screening Visit 1 (Day -35 Visit) and Screening Visit 2 (Day -7 Visit), a negative urine pregnancy test on Day 1, and must not be breastfeeding.
6. Fertile male participants and female participants of childbearing potential must be willing to completely abstain from heterosexual sex or agree to use acceptable contraception from the time of signing informed consent through 30 days after the last dose of study drug.

Exclusion Criteria

1. History of or presence of kidney stones within 1 year prior to Screening.
2. History of or presence of malignancy in the last 5 years other than treated cutaneous basal or squamous cell carcinoma.
3. Hypersensitivity or intolerance to dotinurad or to colchicine and nonsteroidal anti-inflammatory drugs (NSAIDs).
4. Known or suspected history of drug abuse, a positive drug test at Screening Visit 1, or a recent history of alcohol abuse.
5. Known history of or positive results for human immunodeficiency virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV) during Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with an sUA Level <5.0 mg/dL at Week 24 | Week 24

SECONDARY OUTCOMES:
Percentage of Participants who Experience Complete Response (CR) or Partial Response (PR) of ≥1 Target Tophus at Week 76 | Week 76
Percentage of Participants who Experience CR of ≥1 Target Tophus at Week 76 | Week 76
Percentage of Participants with an sUA Level <4.0 mg/dL at Week 24 | Week 24
Mean Rate of Gout Flares Requiring Treatment from Week 36 Through Week 76 | Week 36 through Week 76
Percentage of Participants with an sUA Level <5.0 mg/dL at Week 24 and No Gout Flares Requiring Treatment from Week 36 Through Week 76 | Week 24 and Week 36 through Week 76
Mean Change from Baseline in sUA at Week 24 | Baseline and Week 24
Mean Percent Change from Baseline in the Sum of the Areas for all Target Tophi at Each Visit | Baseline to Week 80
Percentage of Participants who Do Not have a Gout Flare Requiring Treatment from Week 36 through Week 76 | Week 36 through Week 76
Percentage of Participants with an sUA Level <5.0 mg/dL at Each Visit | Up to Week 80
Percentage of Participants with an sUA Level <4.0 mg/dL at Each Visit | Up to Week 80
Percentage of Participants with an sUA Level <3.0 mg/dL at Each Visit | Up to Week 80
Absolute Change from Baseline in sUA Levels at Each Visit | Baseline to Week 80
Percent Change from Baseline in sUA Levels at Each Visit | Baseline to Week 80
Percentage of Participants with a Gout Flare Requiring Treatment at Each Month Between Week 24 and the End of Study | Week 24 to Week 80
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 80
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 80

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates (AARA) - Gilbert, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Associates (AARA) - Glendale, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates (AARA) - Mesa, Mesa, Arizona
  - Del Sol Research Management - Tucson East, Tucson, Arizona
  - Medvin Clinical Research - Covina, Covina, California
  - West Coast Research, Dublin, California
  - Infinity Clinical Research, Norco, California
  - Amicis Research Center - Balboa, Northridge, California
  - Dream Team Clinical Research, Pomona, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - BTC Network - Encompass Clinical Research, Spring Valley, California
  - Cohen Medical Centers, Thousand Oaks, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - Bradenton Research Center, Bradenton, Florida
  - Herco Medical and Research Center, Inc, Coral Gables, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Best Quality Research, Hialeah, Florida
  - Health Awareness Inc, Jupiter, Florida
  - Clinical Research of Center Florida, Lakeland, Florida
  - D&H Pompano Research Center, Margate, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Omega Research DeBary, Orlando, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - DelRicht Research - Atlanta, Atlanta, Georgia
  - Chicago Clinical Research Institute, Inc. (CCRII), Chicago, Illinois
  - Flourish Chicago - Ravenswood (Great Lakes Clinical Trials), Chicago, Illinois
  - MediSphere Medical Research Center, LLC - East, Evansville, Indiana
  - Delricht Research - Better Life Direct Primary Care, Indianapolis, Indiana
  - Delricht Research - Concierge And Direct Primary Care, Overland Park, Kansas
  - DelRicht Research - Louisville (Derby City DPC), Louisville, Kentucky
  - Tandem Clinical Research - Metairie Clinic, Metairie, Louisiana
  - DelRicht Research - LCMC Health Urgent Care - Lakeview, New Orleans, Louisiana
  - DelRicht Research - Prairieville, Prairieville, Louisiana
  - MD Medical Research - Oxon Hill, Oxon Hill, Maryland
  - DelRicht Research - Maryland (Matthew L. Mintz, MD, FACP), Rockville, Maryland
  - MedVadis Research, Waltham, Massachusetts
  - A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Oakland Medical Center, Troy, Michigan
  - Delricht Research - Command Family Medicine, Springfield, Missouri
  - DelRicht Research - Town and Country, Town and Country, Missouri
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Ellipsis Research Group, Brooklyn, New York
  - New York University Langone Orthopedic Center, New York, New York
  - DelRicht Research - Charlotte (Direct Primary Care - DPC), Charlotte, North Carolina
  - Shelby Clinical Research, LLC - North Carolina, Shelby, North Carolina
  - Hometown Urgent Care and Research - Dayton, Dayton, Ohio
  - Delricht Research - Concierge Medicine Of Cincinnati, Mason, Ohio
  - DelRicht Research - Tulsa, Tulsa, Oklahoma
  - Suburban Research Associates - West Chester Office, West Chester, Pennsylvania
  - Coastal Carolina Research Center - Main, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - DelRicht Research - Hendersonville, Hendersonville, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Lone Star Arthritis & Rheumatology Associates - Denton, Denton, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Pioneeer Research Solutions, Houston, Texas
  - Alliance Clinical Lewisville (Epic Clinical Research), Lewisville, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - ERG - Endeavor Clinical Trials, San Antonio, Texas
  - DM Clinical Research - Tomball - Multiple Specialties, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported for publication, after deidentification.
Supporting Information: Study Protocol, SAP